CLINICAL TRIAL: NCT04602403
Title: Does Preoperative Tamsulosin Facilitate Semi-rigid Ureteroscopic Management of Lower Ureteric Calculi Prospective, Randomized Double Blind Study
Brief Title: Does Tamsulosin Facilitate Semi-rigid Ureteroscopic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Ahmed Gaber, Assistant Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: tamsulosin and uretroscopy
Record Dates: First submitted 2020-10-15; First posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Ureter Stone
MeSH Terms: conditions — Ureterolithiasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo group (Placebo Comparator): people who given placebo to become agroup of comparison with the other group
  Interventions: Procedure: rigid ureteroscopy
- tamsulosin group (Active Comparator): people who given tamsulosin to know the effect on ureteroscopy and compare with the control group
  Interventions: Procedure: rigid ureteroscopy

INTERVENTIONS:
Procedure: rigid ureteroscopy — endoscopic treatment of ureteric stones by extraction or peumatic desintegration or laser
  Other Names: endoscopic treatment of ureteric stone

SUMMARY:
Ureteric calculi are one of the most common reasons for frequent Urolithiasis. The estimated prevalence is 8-13% of all calculi.

Medical expulsive therapy (MET) is recommended by the European Association of Urology (EAU) (2013) for 5-10 mm ureteric stones to facilitate stone passage. For MET, alpha blockers, mainly tamsulosin, have shown efficacy in several randomized controlled trials. The underlying pathophysiology of this therapy is supported by the presence and distribution of adrenoreceptors in the ureter. Blocking the action of alpha-1 receptors by pharmacological agents (alpha blockers), such as alfuzosin, terazosin, doxazosin, and, most typically, tamsulosin, results in the relaxation of the ureteric smooth muscle.

Ureteroscopy (URS) is the most commonly performed procedure for the treatment of ureteral calculi, with a high (>90%) stone-free rate after a single treatment. Advancing a rigid ureteroscope into a non-dilated ureter may be difficult and cause complications. Ureteric dilatation may provide access to stones, but not in all cases, and ureteral mucosal injury up to perforation might occur.

DETAILED DESCRIPTION:
Based on the role of alpha blockers, mainly tamsulosin, in MET of ureteric calculus, the investigator will attempt to extend the use of alpha blockers prior to URS for procedural ease. the investigator will conduct a prospective, randomized double-blind study to evaluate whether alpha blockers facilitate the negotiation of the ureteroscope if administered preoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Lower ureteral stone.
* Age: 18 - 75 years.
* normal renal function.
* single sided ureteral stone with normal other kideny.
* sign the informed consent.
* Be willing/able to adhere to follow up visits.

Exclusion Criteria:

* Upper and middle ureteral stones.
* renal impairment.
* Age < 18 years or 75 < years.
* female who were pregnant
* bilateral ureteric stone or solitary kidney.
* urinary tract infection need drainage.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-10-15 (Estimated); Study Completion 2021-10-15 (Estimated)

PRIMARY OUTCOMES:
Rate of patients develop spontaneous expulsion of stone | up to 3 weeks pre operative
  the stone spontaneously expelled without intervension
Number of patients showing dilated ureteric orifice | intraoperative
  during ureteroscopy easy introduction in the ureter
Number of patients need dilatation below stone | intraoperative
  difficult introduce the ureteroscope and reach the stone
Number of patients need dormia extraction or forceps without disintegration | intraoperative
  that is due to dilated ureter so easy remove the stone
Time of operation from introduction of ureteroscope until stone extraction | intraoperative
  to know how easy introduction and expulsion of the ureteroscope

SECONDARY OUTCOMES:
Rate of patients developed side effect from tamsulosin | up to 3 weeks pre operative
  any side effect from alpha blocker
Rate of patients developed complication | intraoperative
  any compliction during ureteroscopy such as perforation
Number of patients show failure of ureteroscopy | intraoperative
  failed introduction or extraction of stone
Number of patients show residual stone post ureteroscopy | postoperative 4 weeks
  difficulty in expulsion of all stones

CONTACTS AND LOCATIONS:
Overall Officials: ahmed m abdel hamed, Study Director — Assiut University
Locations (1):
- Mahmoud Ahmed Gaber, Asyut, Asyut Governorate, Egypt